CLINICAL TRIAL: NCT05056012
Title: Penn Sjögren's International Clinical Collaborative Alliance (SICCA) Follow-up Study
Brief Title: Penn SICCA Follow-up Study
Acronym: PSFS
Status: Not yet recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Vatinee Bunya, MD, Co-Director of Penn Dry Eye & Ocular Surface Center, University of Pennsylvania
Other Study IDs: 827285
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye; Sjogren's Syndrome
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects will provide approximately 7 tablespoons of blood, which may be used for serology, isolation of DNA and isolation of lymphocytes. Subject will have whole saliva sampling performed. These procedures are standardized and validated procedures routinely used for the evaluation of Sjogren's syndrome. Impression cytology may be performed by numbing the ocular surface with drops and then applying a membrane to the conjunctival surface of each eye and the membranes will be stored. A standard Schirmer test will also be performed and strips will be stored after test completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will involve the collection of follow-up data for patients who previously participated in the Sjogren's International Clinical Collaborative Alliance (SICCA) study at the University of Pennsylvania. Clinical data and specimens will be collected from subjects with objective evidence of dry eye who were or were not diagnosed with Sjogren's syndrome at the time of their initial participation in the SICCA study. Specimens will be collected from participants which will include tears, saliva, whole blood, serum, DNA and possible labial minor salivary gland biopsies when indicated. All individuals will participate in a standard evaluation protocol including an oral, ocular and physical examination, objective tests for dry eyes and dry mouth and, whenever necessary, a labial minor salivary gland biopsy. The biopsy requirement is waived for those who have already had positive lip biopsies in the past.

DETAILED DESCRIPTION:
General study design: This is a single center study that involves follow-up of patients who previously participated in the Sjogren's International Collaborative Clinical Alliance (SICCA) at the University of Pennsylvania. Objective evaluation of salivary function will be done by collecting unstimulated whole and stimulated parotid saliva. Objective evaluation of lacrimal function will be performed using the Schirmer test I, Lissamine Green staining, and determining tear break-up time. In a subset of patients, when indicated an objective evaluation of lymphocytic infiltration of the minor salivary glands will be performed by histologic analysis of labial salivary gland biopsies. Serum autoantibody profiles will be determined. In addition, specimens such as biopsies, saliva, sera, conjunctival cells, and tears will be collected. Standardized questionnaires will be used to gain health information.

ELIGIBILITY:
Inclusion Criteria:

1. Previously participated in the SICCA study at Penn
2. Be 18 years or older

4. Have signed an IRB consent form agreeing to the terms of the study

Exclusion Criteria:

1. Did not previously participate in SICCA study at Penn
2. Under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who meet the inclusion/exclusion criteria for this study will be contacted to ask if they would be willing to participate. All recruited participants, who participated in the previous SICCA study at the University of Pennsylvania will be identified.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Collection of specimens and clinical information | 2 years
  To collect specimens (saliva, tears, conjunctival cells, and blood) and clinical information on dry eye patients with or without Sjogren's syndrome

SECONDARY OUTCOMES:
Ocular surface exam findings | 2 years
  Characterize the clinical features of the ocular and oral components of dry eye patients with or without Sjogren's syndrome.
Serologic testing | 2 years
  Characterize the laboratory, including serologic (including autoantibodies), features of dry eye patients with or without Sjogren's syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Vatinee Bunya, MD, Principal Investigator — Scheie Eye Institute
Locations (1):
- Scheie Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided